CLINICAL TRIAL: NCT02383550
Title: Cognitive Evolution in Tysabri Treated Multiple Sclerosis Patients - A Three Year Extension
Acronym: CogMS-Ext
Status: Completed | Type: Observational
Sponsor: Clinique Neuro-Outaouais (Other)
Collaborators: CogState Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNO-002
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational Cognitive assessments — Observational

SUMMARY:
This study is designed to demonstrate that Tysabri is effective in maintaining cognition in MS patients after 5 or more years of continuous treatment.

During a second period of 36 months, the extension study will assess the evolution of cognitive function in Tysabri treated MS patients using the Symbol Digit Modalities Test (SDMT) and a CogState battery of tests.

DETAILED DESCRIPTION:
Tysabri reduces the relapse frequency, slows progression and preserves cognitive function as compared to placebo as per the AFFIRM trial. The benefit on relapse rate and progression appears to be sustained in longer-term studies such as STRATA. In clinical practice however despite a stable EDSS patients often complain of cognitive deterioration.

The investigators' preliminary results from the first pilot study have shown that cognition in Tysabri treated MS patients for two or more years, as measured by the SDMT or Cogstate battery is maintained, including the ability to learn. The investigators' final data will be presented at the American Academy of Neurology (AAN) in 2015.

The Symbol Digit Modalities Test (SDMT) is a sensitive and validated test of cognition in MS. CogState offers a standardized battery of cognitive tests frequently used in clinical research in the fields of dementia and Parkinson's disease. The CogState battery of tests consisting of the Detection test (processing speed), Identification test (attention), One Back test (working memory), International Shopping List test (verbal learning) and the Groton Maze Learning test (reasoning and problem solving) will further confirm and validate the results of the SDMT in MS patients as well as examine other cognitive domains.

The Beck Depression Inventory-II [Beck 1996] is a validated and well recognized clinical research tool for depression in the field of multiple sclerosis.

Together the above tests done prospectively can assess the evolution of cognitive function in Tysabri treated MS patients over the longer term.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the original study and are willing to continue into the extension.

Exclusion Criteria:

* Patients with cognitive decline from causes other than MS (i.e., PML, stroke, sleep apnea, neurodegenerative disorders, brain tumors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis who are receiving Tysabri per indication.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-12; Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
SDMT | 3 years
  Cognitive assessment
Cogstate Battery | 3 years
  Cognitive assessment

CONTACTS AND LOCATIONS:
Overall Officials: Francois Jacques, MD, Principal Investigator — Clinique Neuro-Outaouais
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada